CLINICAL TRIAL: NCT03424031
Title: A Very Early Standing Study in Elderly Stroke
Acronym: AVESSES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Many study exits (many deaths, aggravations) that we had anticipated (but not enough). The patients did not stay long enough in the department to complete the protocol (many study exits that we had not anticipated).
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CHRO-2016-02
Record Dates: First submitted 2018-01-15; First posted 2018-02-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verticalization (Experimental): the patient will be placed in the most vertical position possible.
  Interventions: Procedure: Verticalization
- Passive mobilization (No Intervention): Passive mobilization of the lower limb deficit

INTERVENTIONS:
Procedure: Verticalization — To allow the verticalization of hemiplegic patients, we will use a device commonly used in rehabilitation: the standing (or standing) brand Thera Trainer . This device makes it possible to keep the patient standing despite the motor and postural deficits thanks to knee, buttocks and an anterior support for the upper limbs. Verticalization with this device requires the presence of one or two caregivers (including at least one re-educator), depending on the possibilities of participation of the patient.
  Arms: Verticalization

SUMMARY:
Functional recovery is one of the main issues in the management of stroke and there are various ways in rehabilitation to promote this recovery.

Verticalization is a technique whose benefits have been widely demonstrated, particularly in neurology. Although commonly used in the rehabilitation of stroke, evidence is still lacking as to its impact in this specific care.

Verticalization is underutilized in two situations: in the hyper acute phase as well as in elderly and very deficient patients. It has, however, been shown that the precocity of the treatment allows a better functional recovery. Similarly, the re-education of the elderly is also debated since it has long been mentioned that age was a factor of poor prognosis, the objectives are sometimes underestimated. However, several studies have shown that with the same rehabilitation, elderly patients recover as much as younger patients. The differences found are at least in part due to "less rehabilitation" of older stroke patients.

The different existing data lead us to the hypothesis that the verticalization of the elderly hemiplegic patient in acute phase would allow a better functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* Age > 70
* Modified Rankin Scale (MRS) pre stroke : 0 or 1
* Admission in the neuro vascular unit less than 48 hours after the onset of symptoms
* NIHSS Item 6 for lower extremity motor skills: 3 or 4
* Modified Functional Ambulation Classification : 0
* Affiliated to a social security scheme

Exclusion Criteria:

* History of stroke with motor sequencing limiting walking
* Arterial stenosis limiting the sunrise before D4 (identified by Doppler)
* Symptomatic orthostatic hypotension known or present in the acute phase
* Coma
* Patients who will be referred to a structure (UNV or other) outside the department
* Fracture, orthopedic disorder or any other complication preventing verticalization
* Refusal of the patient to participate in the study or to be verticalized
* Patients under guardianship
* Patients deprived of their liberty by an administrative decision

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
PASS score | 4th month
  the PASS score (score of 36) will be evaluated at 4 months (t2) in single blind (by a physiotherapist who will not be aware of the reeducation performed).

SECONDARY OUTCOMES:
functional recovery | Day 15
  It will be performed in single blind by evaluating the PASS score after the 10th session (t1) or when the patient leaves if it occurs before.
Evaluation of the walk quality | Month 4
  It will be performed in single blind thanks to the modified FAC scale at 4 month
Percentage of days with stools | Day 15
  Number of days with stool / number of days of hospitalization in UNV
Semi-quantitative evaluation | Day 15
  The amount of stool is evaluated in the data collection of the care teams (0: no saddle, +: small amount of stool, ++: moderate amount, +++: larger quantity, ++ ++: very important quantity)

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison R, Dennett R. Pilot randomized controlled trial to assess the impact of additional supported standing practice on functional ability post stroke. Clin Rehabil. 2007 Jul;21(7):614-9. doi: 10.1177/0269215507077364. PMID 17702703
- [Background] Bagg S, Pombo AP, Hopman W. Effect of age on functional outcomes after stroke rehabilitation. Stroke. 2002 Jan;33(1):179-85. doi: 10.1161/hs0102.101224. PMID 11779908
- [Background] Bagley P, Hudson M, Forster A, Smith J, Young J. A randomized trial evaluation of the Oswestry Standing Frame for patients after stroke. Clin Rehabil. 2005 Jun;19(4):354-64. doi: 10.1191/0269215505cr874oa. PMID 15929503
- [Background] Benaim C, Perennou DA, Villy J, Rousseaux M, Pelissier JY. Validation of a standardized assessment of postural control in stroke patients: the Postural Assessment Scale for Stroke Patients (PASS). Stroke. 1999 Sep;30(9):1862-8. doi: 10.1161/01.str.30.9.1862. PMID 10471437